CLINICAL TRIAL: NCT07382869
Title: Impact of Diet and Physical Activity Based Nurse Led Interventions on Maternal Outcome and Neonatal Outcomes in Women With Gestational Diabetes Mellitus (GDM): A Randomized Controlled Trial
Brief Title: to Investigate Impact of Diet and Physical Activity Based Nurse Led Interventions on Maternal Outcomes and Neonatal Outcomes in Women With Gestational Diabetes Mellitus (GDM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Kausar Ghulam Muhammad, MSN Student, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMuhammad
Record Dates: First submitted 2025-12-24; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gestatiaonl Diabetes Mellitus
MeSH Terms: interventions — Walking

STUDY DESIGN:
Intervention Model Description: Diet plan, Arm chair Exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: Standard Care (No Intervention): Participants in the control group will receive standard care.
- Experimental group (Experimental): Experimental group will receive nurse led intervention including diet,arm chair exercise and walk.
  Interventions: Other: Arm chair exercise, Walk, Diet plan will be given to experimental group.

INTERVENTIONS:
Other: Arm chair exercise, Walk, Diet plan will be given to experimental group. — Participants in the intervention group will receive nursing intervention sessions by researcher focusing on:
  * Dietary modifications based on caloric needs and glycemic index education.
  * Safe physical activity such as walk for 150 minutes per week (30 minutes daily).
  * Physical exercise under supervision of nurse physical activity guidance.
  * To assess in the management of gestational diabetes mellitus participants will be instructed to perform simple arm raises exercise using light weights. Each session will be scheduled for 10-15 minutes and conducted three times per weeks to promote upper body strength. Studied suggest that resistant training for 20 -30 minutes a week can reduce insulin resistance. The exercise regimen will be structured to incorporate these recommendations. Participants in the active arm exercise received written step prescriptions, and set individualized targets (Diabetes Canada, 2025).
  * Follow-up on alternate week (15 days) and 5 counseling sessio
  Arms: Experimental group

SUMMARY:
Gestational Diabetes Mellitus (GDM) is a growing maternal health concern associated with adverse neonatal outcomes such as macrosomia and shoulder dystocia, often aggravated by poor dietary habits and physical inactivity during pregnancy. This randomized controlled study aims to evaluate the effectiveness of structured nursing interventions focusing on diet and physical activity in improving maternal glycemic control and reducing neonatal complications. A total of 66 pregnant women diagnosed with GDM will be selected through purposive sampling and randomly allocated into intervention and control groups using the lottery method. The intervention group will receive individualized dietary counselling, pregnancy-appropriate physical activity guidance, and regular nursing follow-up, while the control group will continue with routine antenatal care. Maternal outcomes, including fasting blood glucose and HbA1c levels, will be measured at baseline and follow-up visits. Neonatal outcomes such as macrosomia, mode of delivery, and shoulder dystocia will be documented at birth. Data will be collected using structured tools and analysed using SPSS, with independent t-tests and chi-square tests applied. The study anticipates that structured nursing interventions will significantly improve glycaemic control and reduce adverse neonatal outcomes, supporting the integration of evidence-based nursing care into routine GDM management.

DETAILED DESCRIPTION:
Gestational Diabetes Mellitus (GDM) is a growing concern in maternal health, often leading to complications like macrosomia and shoulder dystocia that affect neonatal outcomes. Poor dietary habits and sedentary lifestyles during pregnancy further worsen glycemic control in women with GDM. This study aims to evaluate the impact of structured nursing interventions focused on diet and physical activity on maternal blood sugar levels and neonatal outcomes, particularly macrosomia and shoulder dystocia. The research will test the hypothesis that diet and physical activity-based nursing interventions significantly improve glycemic control and reduce the risk of adverse neonatal outcomes compared to routine prenatal care. The main objectives are to assess changes in maternal fasting blood glucose and HbA1c levels and to evaluate the incidence of macrosomia and shoulder dystocia in neonates. This randomized controlled study will be conducted among 66 pregnant women diagnosed with GDM. Participants will be selected using purposive sampling and assigned to either the intervention group or control group using lottery methods. The intervention group will receive personalized nursing support, including diet education, physical activity guidance tailored for pregnancy, and regular follow-up, while the control group will continue with standard antenatal care. Maternal parameters such as fasting blood glucose, and HbA1c levels will be recorded at baseline and during follow-up visits.

Neonatal outcomes, including macrosomia, mode of delivery, and presence of shoulder dystocia, will be documented at delivery. All data will be collected by the researcher using structured data collection tools. Statistical analysis will be performed using SPSS. Descriptive statistics will summarize demographics and baseline data. Independent t-tests will compare glycaemic outcomes; chi-square tests will be used to compare neonatal outcomes. The anticipated outcome is that diet and physical activity-based nursing interventions will lead to improved maternal glycaemic control and significantly reduce neonatal complications. This study may offer evidence supporting the integration of structured nursing care into routine gestational diabetes mellitus management and this also contribute toward the betterment in terms of maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18-40 years

* Diagnosed with GDM in the indexed pregnancy
* Singleton pregnancy. Pregnant women with gravida 02.

Exclusion Criteria:

* Pre-existing diabetes mellitus (Type 1 or Type 2)
* Multiple pregnancies (twins, triplets, etc.)
* Women with history of Pregnancy induced hypertension. (PIH)
* History of chronic medical conditions (renal disease, cardiac disorders, epilepsy)
* Psychiatric illness or cognitive impairment that may affect participation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females with indexed gestational diabetes millitus.
Enrollment: 66 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maternal glycemic control assessed by HbA1c (%) | Baseline (at enrollment: 24-28 weeks gestation) to 36-38 weeks gestation
  Change in maternal glycemic control measured by glycated hemoglobin (HbA1c, %) using standardized laboratory blood assays from baseline (at enrollment) to 36-38 weeks of gestation.
Fasting plasma glucose (mg/dL) | Baseline (24-28 weeks gestation) to 36-38 weeks gestation
  Change in fasting plasma glucose levels (mg/dL) measured using a fasting venous blood sample at baseline and at 36-38 weeks of gestation.

SECONDARY OUTCOMES:
Mode of delivery | Mode of delivery (vaginal or cesarean section) recorded from hospital obstetric records at the time of childbirth.
  At delivery
Neonatal birth weight (grams) | Neonatal birth weight (grams) measured within the first hour after birth using a calibrated neonatal weighing scale.
  At birth
Neonatal Apgar score | Apgar score assessed at 1 and 5 minutes after delivery using the standard Apgar scoring system.
  1 minute and 5 minutes after birth
Neonatal complications | Incidence of neonatal complications, including shoulder dystocia and neonatal hypoglycemia, assessed through standard clinical examination and review of neonatal medical records within 48 hours after birth.
  From birth to 48 hours postpartum
Secondary Outcome Measure 5 | Description: Maternal weight change measured in kilograms (kg) from enrollment to delivery using routine antenatal weight records.
  Title: Gestational weight gain (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lamia Yusuf, FCPS, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University Of Health Sciences,Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brown J, Ceysens G, Boulvain M. Exercise for pregnant women with pre-existing diabetes for improving maternal and fetal outcomes. Cochrane Database Syst Rev. 2017 Dec 21;12(12):CD012696. doi: 10.1002/14651858.CD012696.pub2. PMID 29264871
- See also: Article:Effects of comprehensive nursing intervention on maternal and infant outcomes for gestational diabetes mellitus patients — https://link.springer.com/article/10.1007/s13410-020-00816-5#citeas